CLINICAL TRIAL: NCT02809638
Title: Ultrasound Elastography: a New Technique to Diagnose Acute and Chronic Deep Vein Thrombosis
Brief Title: A New Technique to Diagnose Acute and Chronic Deep Vein Thrombosis
Status: Completed | Type: Observational
Sponsor: Azienda Sanitaria Locale ASL 6, Livorno (Other Government)
Responsible Party: Principal Investigator, Nicola Mumoli, Azienda Sanitaria Locale ASL 6, Livorno, Azienda Sanitaria Locale ASL 6, Livorno
Other Study IDs: Azienda USL Toscana Nord Ovest
Record Dates: First submitted 2016-05-30; First posted 2016-06-22 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Deep Vein Thrombosis; Compression Ultrasound; Elastography; Elasticity Imaging Techniques
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DVT of the lower limbs: patients with first suspected episode of unprovoked DVT of the lower limbs and patients with episode of unprovoked DVT of the lower limbs at third month of follow-up
  Interventions: Other: ultrasound elastography

INTERVENTIONS:
Other: ultrasound elastography

SUMMARY:
In clinical practice, compression ultrasound (CUS) has become an easy and reliable noninvasive tool for the diagnosis of deep vein thrombosis (DVT).

Currently there are not validated methods to assess the biological age of venous thrombus, and the date of onset of thrombosis. One potential technique to age DVT is ultrasound elastography (UE). UE is a noninvasive technique to measure tissue hardness, and it is well known that thrombi harden as they age. The aim of this study will be to assess the ability of UE to distinguish acute from chronic DVT. The investigators will evaluate prospectively all consecutive outpatients presenting with clinically suspected unprovoked DVT of the lower limbs, and those having a previous diagnosis of DVT for the scheduled 3 months visit of follow-up, for a period of about one year. All the enrolled patients will undergo to the CUS of the lower limbs, and at the same time to the ultrasound elastography by the physician expert in vascular ultrasound. The specialist performing both examinations will be unaware of the time of onset of DVT (acute or chronic). Then the patients will be divided into two groups (group A: patients with acute DVT; group B: patients with chronic DVT at the 3rd month of follow-up). Each examination (CUS and ultrasound elastography) will be repeated three times in the same patient at the same visit, to assess the reproducibility of the technique. The demographic data, medical history, physical examination and the results of CUS and ultrasound elastography will be collected in a case report form (CRF) by another investigator who does not perform the examinations. The blinded CRF will be submitted to a dedicated committee for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* acute first episode of unprovoked DVT of lower limbs
* chronic first episode of unprovoked DVT of lower limbs (at third month of follow up)

Exclusion Criteria:

* previous episodes of DVT
* ongoing anticoagulation
* age younger than 18 years
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this study, we will evaluate prospectively all consecutive outpatients presenting with clinically suspected unprovoked DVT of the lower limbs, and those having a previous diagnosis of DVT for the scheduled 3 months visit of follow-up, for a period of about one year. All the enrolled patients will undergo to the CUS of the lower limbs, and at the same time to the ultrasound elastography by the physician expert in vascular ultrasound. The specialist performing both examinations will be unaware of the time of onset of DVT (acute or chronic). Then the patients will be divided into two groups (group A: patients with acute DVT; group B: patients with chronic DVT at the 3rd month of follow-up). Each examination (CUS and ultrasound elastography) will be repeated three times in the same patient at the same visit, to assess the reproducibility of the technique.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-08; Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

PRIMARY OUTCOMES:
Density of clots in patients having acute or 3 month DVT of the lower limb, using the technique of elastosonography. | 1 year

SECONDARY OUTCOMES:
Change of the density of the clots measured by elastosonography, assessing the elastic deformability of the thrombus, and correlating it with the time of occurrence of the thrombosis (fresh or three month aged clots) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Mumoli, M.D., Study Chair — Department of Internal Medicine, Livorno Hospital, Livorno, Italy
Locations (1):
- Azienda USL 6 Livorno, Livorno, Tuscany, Italy